CLINICAL TRIAL: NCT04334837
Title: An Open-Label, Multi-Center Expanded Access Protocol of Copper Cu 64 Dotatate for the Detection, Localization and Monitoring of Somatostatin Receptor Expressing Neuroendocrine Tumors (NETs)
Brief Title: Copper Cu 64 Dotatate for the Detection, Localization and Monitoring of SSTR Expressing (NETs)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Curium US LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CURCu64Dot0001
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Neuroendocrine Tumors
Keywords: Somatostatin; 64Cu-DOTATATE; Neuroendocrine; PET/CT; PET/CT in oncology; Radiopharmaceuticals; Cu-64; Copper-64
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Diagnostic Test: Copper Cu 64 Dotatate — The drug product contains Copper Cu 64 Dotatate filled in a glass vial, closed with butyl rubber stopper secured with an aluminum crimp seal. The drug product will be delivered by Curium to the clinical site. The EAP drug will be administered as an intravenous bolus injection. The dose will be administered according to the schedule detailed in the protocol.

SUMMARY:
This is an open-label, multi-center expanded access program designed to provide access to Copper Cu 64 Dotatate for the detection, localization, and monitoring of NETs to patients that did not have access during the Phase 3 Trial.

DETAILED DESCRIPTION:
The objective of this trial is to provide patients with confirmed or suspicion of NET access to Copper Cu 64 Dotatate for the detection, localization, and monitoring of SSTR expressing NETs, bridging the gap between investigational product availability in clinical studies and marketed product availability following US Food and Drug Administration (FDA) approval.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, aged ≥18 years.
* Willing to sign the Informed Consent Form.
* Able to understand and comply with the procedures and requirements of the program.
* Meet at least one of the following criteria:

  1. Confirmed or suspicion of NET based on histology/biopsy report.
  2. Confirmed or suspicion of NET based on conventional imaging scans of affected area such as MRI and/or contrast enhanced CT and/or an FDG PET-CT scan and/or NaF PET-CT scan and/or OctreoScan® and/or clinical symptoms performed within 8 weeks prior to administration of Copper Cu 64 Dotatate.
* Negative pregnancy test in women of child-bearing potential, using urine (dip stick test) or blood based testing (within 48 hours of injection).
* For women of childbearing potential, agreement to remain abstinent (refrain from heterosexual intercourse) or use non-hormonal contraceptive methods for at least 2 weeks following administration of investigational product.
* For men, agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures for at least 2 weeks following administration of investigational product.
* Recent blood test results (within 4 weeks pre-dose) as follows:

  1. WBC: >2 x 109/L
  2. Hemoglobin: >8.0g/dL
  3. Platelets: >50 x 109/L
  4. ALT, AST, AP: ≤5 times ULN
  5. Bilirubin: ≤3 times ULN
  6. Serum creatinine: <170 μmol/L

Exclusion Criteria:

* Pregnant, planning to be pregnant within the next two weeks.
* Therapeutic use of any somatostatin analogue, including Sandostatin® LAR and Lanreotide (within 28 days) and Sandostatin® (within 2 days) prior to administration with Copper Cu 64 Dotatate. If a patient is on Sandostatin® LAR or Lanreotide, a wash-out period of 28 days is required before the injection of the investigational product.
* History or presence of significant hematological abnormalities or immunodeficiency or any condition that might compromise the immune system (infections, vaccinations), of any etiology as indicated by clinically significantly abnormal values of any of the following hematologic parameters: platelets, hemoglobin, WBC count and ANC.
* Lactating and breast-feeding women.
* Acute or chronic clinically significant conditions such as uncontrolled congestive heart failure (rule out with MUGA scan, if suspected), liver or kidney dysfunction, uncontrolled hypertension.
* History of hypersensitivity to drugs with a similar chemical structure to the investigational product or any of its excipients.
* History of significant drug abuse within 1 year prior to administration of Copper Cu 64 Dotatate. Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine, and crack) within 1 year prior to administration of Copper Cu 64 Dotatate.
* Participation in other clinical research trials involving evaluation of other investigational treatments within 30 days prior to administration of Copper Cu 64 Dotatate and/or unwilling to allow at least one week before participation in another drug trial following administration of Copper Cu 64 Dotatate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult